CLINICAL TRIAL: NCT01944956
Title: Swallow Maturation in Preterm and Term Infants
Brief Title: Swallowing Sound in Preterm Infant Evaluation of Feeding Maturation
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Deniz Anuk Ince, Principal Investigator, Baskent University
Other Study IDs: Baskent; swallowing sounds preterm (Registry Identifier: swallowing sounds preterm infants); Deniz (Registry Identifier: Deniz)
Record Dates: First submitted 2013-09-11; First posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2011-03

CONDITIONS: Other Preterm Infants
Keywords: Maturation; preterm infants; sucking and swallowing

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Our objective was to evaluate maturation of sucking and swallowing in preterm infants using a non-invasive method: assessment of swallowing sounds. Findings in healthy term infants were used as reference values.

DETAILED DESCRIPTION:
Successful transition to full oral feeding in preterm infants is important for safe discharge from hospital and for facilitating the mother-infant bond. Preterm infants were evaluated weekly for sucking and swallowing performance (i.e., feeding performance) from the time they began oral feeding (frequency 1-2 oral feedings/day) until they reached independent oral feeding (frequency 8 oral feedings/day) at postmenstrual 38-40 weeks. For the term infants, we evaluated a single oral feeding during the first week of life.

The exclusion criteria were major congenital abnormalities, craniofacial malformation, intracranial hemorrhage, bronchopulmonary dysplasia, culture-positive sepsis, and necrotizing enterocolitis. Each swallowing-sound recording was 2 minutes long and was captured in a quiet environment by the same investigator. The feeding parameters generated from the recordings were as follows: total number of swallows (S), total number of rhythmic swallows (RS), total number of resting intervals (RI), average time between resting intervals (ATRI), average time between swallows (ATS), average time between rhythmic swallows (ATRS), maximum number of rythymic swallows (MRS), and volume of milk ingested (VM) during the 2-minute evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants (< 37 gestational weeks) and term infants (>=37 gestational weeks)

Exclusion Criteria:

- The exclusion criteria were major congenital abnormalities, craniofacial malformation, intracranial hemorrhage, bronchopulmonary dysplasia, culture-positive sepsis, and necrotizing enterocolitis.

Ages: 26 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants (< 37 gestational weeks) and term infants (>=37 gestational weeks)
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
swallow count | Participants will be followed up until postmenstrual 38-40 weeks, an expected avarage of 10 weeks
  Mean MRS (mean±SD;17±7) for the preterm group reached the reference value at postmenstrual 38-40 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Anuk Ince, MD, Principal Investigator — Baskent University

REFERENCES:
- [Derived] Ince DA, Ecevit A, Acar BO, Saracoglu A, Kurt A, Tekindal MA, Tarcan A. Noninvasive evaluation of swallowing sound is an effective way of diagnosing feeding maturation in newborn infants. Acta Paediatr. 2014 Aug;103(8):e340-8. doi: 10.1111/apa.12686. Epub 2014 May 29. PMID 24814215